CLINICAL TRIAL: NCT06138249
Title: Different Kinds of Vitamin D Intake and Its Metabolites: Blood Levels and Bone Mineral Density. A Randomized Clinical Trial.
Brief Title: Cholecalciferol and Calcifediol Are Both Useful to Improve Vitamin D Serum Levels
Acronym: VITD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Silvana De Giorgi (Unknown); Davide Bizzoca (Unknown); Angela Notarnicola (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VITD
Record Dates: First submitted 2023-07-21; First posted 2023-11-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcifediol each month (Experimental): Calcifediol 0,266 mg each month
  Interventions: Dietary Supplement: Vitamin D
- Cholecalciferol 25.000 UI (Experimental): Cholecalciferol 25000UI each 15 days
  Interventions: Dietary Supplement: Vitamin D
- Calcifediol 4 drops each day (Experimental): Calcifediol 4 drops each day
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D

SUMMARY:
Patients with hypovitaminosis D are randomized into three arms of treatment:

Group A: Calcifediol 0,266mg each month Group B: Cholecalciferol 25000UI each 15 days Group C: Calcifediol 4 drops per day. Serum levels of vitamin D are dosed after one month of treatment

DETAILED DESCRIPTION:
Patients with hypovitaminosis D are randomized into three arms of treatment:

Group A: Calcifediol 0,266mg each month Group B: Cholecalciferol 25000UI each 15 days Group C: Calcifediol 4 drops per day. Serum levels of vitamin D are dosed after one month of treatment to support the best dosage of Vitamin D intake.

ELIGIBILITY:
Inclusion Criteria:

* Hypovitaminosis D (<20ng/mL)

Exclusion Criteria:

* Osteoporosis (T score <-2.5SD)
* Renal or hepatic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
level of Vitamin D | Between recruitment and 1 month
  Blood dosage of Vitamin D
level of Vitamin D | Between recruitment and 6 month
  Blood dosage of vitamin D

SECONDARY OUTCOMES:
DEXA | Between recruitment and 18 months
  DEXA is a radiographic measurement of Bone Mass

CONTACTS AND LOCATIONS:
Overall Officials: Angela Notarnicola, AP, Study Chair — University of Bari
Locations (1):
- University of Bari, Bari, Italy

REFERENCES:
- [Background] Paterson C. Vitamin D deficiency: a diagnosis often missed. Br J Hosp Med (Lond). 2011 Aug;72(8):456-8, 460-2. doi: 10.12968/hmed.2011.72.8.456. PMID 21841591
- [Background] Castano L, Madariaga L, Grau G, Garcia-Castano A. 25(OH)Vitamin D Deficiency and Calcifediol Treatment in Pediatrics. Nutrients. 2022 Apr 29;14(9):1854. doi: 10.3390/nu14091854. PMID 35565821
- [Background] Haddow JE. Vitamin D and rickets: much has been accomplished, but there is room for improvement. J Med Screen. 2011;18(2):58-9. doi: 10.1258/jms.2011.011059. No abstract available. PMID 21852696
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/